CLINICAL TRIAL: NCT01471431
Title: A Randomized Trial of the Spontaneous Breathing Trial to Extubate Very Low Birthweight Infants
Brief Title: Extubation Readiness Study in Very Low Birthweight Infants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility analysis by DSMC recommended termination.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 813859
Record Dates: First submitted 2011-11-10; First posted 2011-11-16 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2015-09

CONDITIONS: Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spontaneous breathing trial (Experimental): The spontaneous breathing trial will determine the extubation readiness of the subject.
  Interventions: Other: spontaneous breathing trial
- Usual care (No Intervention): Subjects will be extubated using usual care, without the use of the spontaneous breathing trial.

INTERVENTIONS:
Other: spontaneous breathing trial — The SBT is performed daily on rounds if an infant is on conventional ventilation and meets all predetermined ventilator criteria (set ventilator rate ≤30, peak inspiratory pressure (PIP) delivered on mandatory breaths ≤20 cm H2O, pressure support (PS) ≤8 cm H2O, positive end-expiratory pressure (PEEP) ≤6 cm H2O, inspired fractional oxygen (FiO2) ≤0.40).
  During the SBT, the ventilator rate and pressure support are set to zero, and the infant is maintained on continuous positive airway pressure (CPAP) alone via the endotracheal tube. The trial duration is 3 minutes, unless an infant fails before the trial is complete. Failure is defined as bradycardia <100 for >15 seconds or oxygen saturation by pulse oximetry <85% despite a 15% increase in FiO2. If an infant passes the SBT, they are extubated within 3 hours. If an infant fails the SBT, they remain intubated and the daily application of the SBT continues as long as the minimum ventilator criteria are met.
  Arms: Spontaneous breathing trial

SUMMARY:
The objective of this study is to determine whether use of the spontaneous breathing trial allows for earlier successful extubation of very low birth weight (VLBW) infants who are intubated for >48 hours and have not yet been successfully extubated (extubated >7 days).

ELIGIBILITY:
Inclusion Criteria:

* Birthweight >500g and<1500g.
* Postmenstrual age <34 weeks
* Mechanically ventilated >48 hours
* Never successfully extubated

Exclusion Criteria:

* Congenital heart disease (other than patent ductus arteriosus (PDA), patent foramen ovale (PFO), and restrictive ventricular septal defect (VSD)
* Known or suspected airway anomalies
* Severe congenital malformations
* Need to remain intubated for other reasons (i.e. having surgery)
* Has met SBT criteria on previous calendar day (after 48 hrs of ventilation, PIP≤18, PEEP≤6, FiO2≤40%, Rate≤30, PS≤8)

Ages: 48 Hours to 14 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2011-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
time to successful extubation | 34 weeks postmenstrual age
  The time from intubation (if >48 hours) to successful extubation (if > 7 days) as evaluated at 34 weeks postmenstrual age (gestational age + chronologic age)

SECONDARY OUTCOMES:
bronchopulmonary dysplasia | 36 weeks postmenstrual age
  The diagnosis of bronchopulmonary dysplasia will be made at 36 weeks postmenstrual age, using the traditional definition and the NIH Consensus definition.
extubation failure rate | 34 weeks postmenstrual age
  The proportion of infants who fail extubation will be compared between the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Johanna Giaccone, MD, Study Director — University of Pennsylvania; Barbara Schmidt, MD, MSc, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - The Hospital of the University of Pennsylvania, Phialdelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania